CLINICAL TRIAL: NCT05802147
Title: Analyse Of Early Skın To Skın Contact's Impact Upon Maternal-Infant Bondıng And Perceptıon Of Traumatıc Bırth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Okçu, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10436591
Record Dates: First submitted 2023-01-29; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Postpartum
Keywords: traumatic birth; maternal attachment; Skin to skin; Midwifery
MeSH Terms: conditions — Birth Injuries

STUDY DESIGN:
Intervention Model Description: This study was carried out as a randomized controlled experimental study in order to examine the effect of early skin-to-skin contact on mother-infant attachment and traumatic birth perception and to provide new information to the literature. The sample of the study consisted of 350 women who applied to the Training and Research Hospital in the city center of Batman between December 2021 and May 2022, and who agreed to participate as the study group (n: 175) and the control group (n: 175), who had a normal delivery in the delivery room has created.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Skin to Skin Contact Group (Experimental): Women who met the criteria for inclusion in the study and accepted the study (n:180) were told how to apply skin-to-skin contact. Skin-to-skin contact was initiated within the first minutes of normal delivery and skin-to-skin contact was applied to the mothers for a minimum of 15 minutes (due to the high number and frequency of births in the TDL service and hospital conditions). Routine newborn care procedures (eye drops, vaccination, footprints, etc.) performed in the delivery room were performed during skin-to-skin contact. After the skin-to-skin contact between the mother and the newborn was terminated at the end of delivery, 2 hours later, mothers were asked to fill in a personal questionnaire and a traumatic birth scale. The maternal attachment scale was completed 1 month after birth by telephone interview.
  Interventions: Behavioral: skin-to-skin contact
- Control Group (No Intervention): Standard midwifery practices and labor follow-up were applied to women who met the inclusion criteria in the hospital (during the delivery room) (n: 187), agreed to participate in the study, and were in the control group. Neonatal routine care procedures (vaccine, footprint, eye drop application, etc.) of the postpartum hospital were performed. Then, after 2 hours postpartum, mothers were asked to fill in a personal questionnaire and a traumatic birth scale. The maternal attachment scale was completed 1 month after birth by telephone interview.

INTERVENTIONS:
Behavioral: skin-to-skin contact — skin-to-skin contact
  Arms: Early Skin to Skin Contact Group

SUMMARY:
This study will carry out as a randomized controlled experimental study in order to examine the effect of early skin-to-skin contact on mother-infant attachment and traumatic birth perception and to provide new information to the literature. The sample of the study consist of 350 women who apply to the Training and Research Hospital in the city center of Batman between December 2021 and May 2022, and who agreed to participate as the study group (n:175) and the control group (n: 175), who had a normal delivery in the delivery room. hascreated. "Personal Questionnaire Form", "Traumatic Birth Perception Scale" and "MaternalAttachment Scale" forms were used in the analysis of the data. Data analysis was done with SPSS 24 program

DETAILED DESCRIPTION:
The population of the study consisted of puerperant women who gave normal birth in Batman Training and Research Hospital TDL (Travay-Birth-Postpartum) service between December 2021 and May 2022. The population of the research was determined as N:2760 for the 6-month data collection period in the center with a monthly average of 460 normal births.The sample of the study consisted of women who met the research conditions and accepted the study. In our study, the sample population was calculated as n:338 people with a 95% confidence interval using the known sample calculation method. The sample number was determined as n:367 puerperant women, since there may be a loss of cases in the research (desire to leave the research, interruption of attachment, not filling out the entire questionnaire…).

Inclusion Criteria: Agreeing to participate in the study, Vaginal delivery, Being between 37-42 weeks of gestation, Hearing and visual impairment, Be between 18-49 years old, No psychiatric diagnosis, Reading and writing Turkish and understanding Turkish, Single and healthy fetus, Head presentation, Not having a high-risk pregnancy, No need for neonatal intensive care Exclusion Criteria in Research: Not meeting the inclusion criteria,Not completing the forms, Multiple pregnancy, Women who refused to participate in the study were excluded from the study.

Randomization: In order to keep the number of people in balance between the groups, the "block randomization" method, one of the fixed-probability randomization methods, was used. By using a computer program module (http://www.randomr.org/form.htm) used in randomization-controlled studies using the block randomization method, the data were collected at one-week intervals considering the inclusion criteria in order not to affect the groups compared to each other. group (A), 2nd week control group (B), 3rd week study group (A), 4th week control group (B), …)." Which group to start with first was determined by a person independent of the research using the coin-print method.

Working Group: Women who met the criteria for inclusion in the study and accepted the study (n:180) were told how to apply skin-to-skin contact. Skin-to-skin contact was initiated within the first minutes of normal delivery and skin-to-skin contact was applied to the mothers for a minimum of 15 minutes (due to the high number and frequency of births in the TDL service and hospital conditions). Routine newborn care procedures (eye drops, vaccination, footprints, etc.) performed in the delivery room were performed during skin-to-skin contact. After the skin-to-skin contact between the mother and the newborn was terminated at the end of delivery, 2 hours later, mothers were asked to fill in a personal questionnaire and a traumatic birth scale. The maternal attachment scale was completed 1 month after birth by telephone interview.

Control Group: Standard midwifery practices and labor follow-up were applied to women who met the inclusion criteria in the hospital (during the delivery room) (n: 187), agreed to participate in the study, and were in the control group. Neonatal routine care procedures (vaccine, footprint, eye drop application, etc.) of the postpartum hospital were performed. Then, after 2 hours postpartum, mothers were asked to fill in a personal questionnaire and a traumatic birth scale. The maternal attachment scale was completed 1 month after birth by telephone interview

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study
* Do not give vaginal birth
* Being between 37-42 weeks of gestation
* Not having a hearing or visual impairment
* Being between the ages of 18-49
* Not having a psychiatric diagnosis
* Reading and writing Turkish and understanding Turkish
* Single and healthy fetus
* Chief presentation
* Not having a risky pregnancy
* No need for neonatal intensive care

Exclusion Criteria:

* Not meeting the inclusion criteria,
* Not completing the forms,
* Having multiple pregnancy,
* Women who refused to participate in the study were excluded from the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 350 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Maternal Attachment Scale Score | from birth to 1 month after birth
  Maternal attachment scale, developed by Mary E. Muller in 1994 and adapted to Turkish by Kavlak and Şirin in 2009, was used to evaluate the bond between mother and baby.
Traumatic Birth Perception Scale Score | from birth up to 2 hours after birth
  It was evaluated with the Traumatic birth perception scale developed by Yalnız et al. (2016) to determine the perception of traumatic birth.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatice OKÇU, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No